CLINICAL TRIAL: NCT05279599
Title: Application of Circulating Extracellular Vesicles in Early Disease Assessment and Prognosis After Traumatic Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TDSJWKTBIEX
Record Dates: First submitted 2022-01-26; First posted 2022-03-15 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Traumatic Brain Injury
Keywords: molecular markers; prognosis; inflammation; peripheral circulation
MeSH Terms: conditions — Brain Injuries, Traumatic; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Peripheral blood was collected in a negative pressure vacuum tube and transferred to the refrigerator -80 for storage as soon as possible.
  2. Peripheral blood-related cells are subsequently collected or cultured to observe the relationship between related molecules and circulating extracellular vesicles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study was to observe the relationship between the changes of circulating extracellular vesicles and disease development and outcome in patients with traumatic brain injury, and to find early serum markers and potential intervention targets for disease monitoring in patients with traumatic brain injury. In addition, explore the source of extracellular vesicles as much as possible to prepare for subsequent basic experiments.

DETAILED DESCRIPTION:
To compare the changes of molecular markers and circulating-related cell phenotype molecules in the serum of patients with traumatic brain injury, to observe the relationship between the changes of circulating extracellular vesicles and the development and outcome of the disease in patients with traumatic brain injury, and to search for early serum markers of patients with traumatic brain injury and potential interventions.

ELIGIBILITY:
Inclusion Criteria:

1. No systematic treatment before admission;
2. The patient is diagnosed with traumatic brain injury with imaging evidence;
3. Age > 18 years old;
4. The patient or family members agree to sign the informed consent.

Exclusion Criteria:

1. Infectious diseases within the past 1 month;
2. Past head trauma, history of neurological diseases;
3. Non-isolated traumatic brain injury;
4. The patient is not receiving treatment in this hospital;
5. Severe disability, dementia, or organ dysfunction before the onset of the disease;
6. Subject refuses to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All TBI patients treated at Tangdu Hospital from January 2022 to December 2022
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
The type and content of circulating extracellular vesicles | within 24 hours of TBI
  After isolation of circulating extracellular vesicles, RNA sequencing was performed to determine noncoding RNA changes in circulating extracellular vesicles. Screening criteria were based on logFC and P value, generally with |logFC|>2 and AP value <0.05 to define whether there was a difference.
Neurological deterioration in patients with traumatic brain injury | within 7 days after injury
  Neurological deterioration (ND) was defined as the occurrence of one or more of the following criteria within 7 days after injury: (a) a decrease in GCS score of 2 points or more from the initial GCS score with no pharmacological sedation; (b) a deterioration in neurological status being sufficient to neurosurgical intervention.

SECONDARY OUTCOMES:
hospital stay | From hospitalization to discharge，up to one month
  The cumulative number of days from admission to discharge of the patient. Regardless of whether the admission and discharge were in the morning or afternoon, the total admission and discharge was one day. It mainly reflects the turnover of hospital beds.
GOSE score | three months or six months
  The GOSE score was dichotomized into being moderately disabled or worse (GOSE score ≤6) versus good recovery (GOSE score 7-8), and into being severely disabled or worse (GOSE score ≤4) versus moderate or no disability (GOSE score 5-8).

CONTACTS AND LOCATIONS:
Overall Officials: Yan Qu, M.D, Ph.D, Study Chair — Tang-Du Hospital; Qing Hu, M.D, Principal Investigator — Tang-Du Hospital
Locations (1):
- Tandu Hospital, Fourth Military Medical University, Xi'an, China